CLINICAL TRIAL: NCT05469594
Title: Second-trimester Termination of Pregnancy: A Retrospective Study Comparing Complications Related to Termination of Pregnancy at 12-14 Weeks' Gestation Versus 14-16 Weeks' Gestation
Brief Title: Second-trimester TOP : a Retrospective Study Comparing Complications at 12-14 vs 14-16 Weeks of Gestation
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Kevin GUILLEZ, Specialist assistant in gynaecology and obstetrics, Central Hospital, Nancy, France
Other Study IDs: 2022PI033-230
Record Dates: First submitted 2022-07-11; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Abortion in First Trimester; Abortion, Second Trimester
Keywords: complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Termination of pregnancy between 12-14 weeks of gestation
- Termination of pregnancy between 14-16 weeks of gestation

SUMMARY:
In France, the recently adopted law relating to the legal time limit for access to voluntary interruption of pregnancy has set a threshold of the term at which it can be performed up to 16 weeks of gestation. This single-centre study conduced at the Nancy Maternity Hospital is based on a retrospective cohort of all patients who underwent a medical termination of pregnancy between January 2010 and October 2021. The main objective is to evaluate the complications according to the term of the termination of pregnancy between two groups : [12-14] vs [14-16] weeks of gestation. The secondary objective is the distribution of these complications between the two groups. Pregnancy termination can be performed in two methods, either by medical method with mifepristone and misoprostol, or by surgical method by dilation and evacuation. Complications identified are haemorrhage, infection, retained product of trophoblast, uterine rupture and abortion induction failure. The hypothesis is the concomitant increase in complications with the term of the termination of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* termination of pregnancy for a medical reason
* between 12 and 16 weeks of gestation
* singleton pregnancy

Exclusion Criteria:

* multiple pregnancy
* abortion occurred before the induction of termination of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women of childbearing age, major, with a single pregnancy who underwent for termination of pregnancy for medical reasons (maternal or foetal) between 12 and 16 weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
complications | Day 0
  hemorrhage, infection, retained product of conception, failure, uterine rupture

SECONDARY OUTCOMES:
repartition of all complications | Day 0
  repartition of all complications between groups